CLINICAL TRIAL: NCT03829995
Title: Effect of Pharmacist Provided Drug Information Services After Hospital Discharge: Patient Satisfaction and Sense Of Security Regarding Drug Treatment.
Brief Title: Effect of Pharmacist Provided Drug Information Services After Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Hovedstadens Apotek (Other Government)
Collaborators: The Hospitals Pharmacies' and Amgros' Research Development Foundation (Unknown)
Responsible Party: Principal Investigator, Tim Emil Vejborg, Principal Investigator, Region Hovedstadens Apotek
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-18003889
Record Dates: First submitted 2019-01-22; First posted 2019-02-04 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Drug Counseling

STUDY DESIGN:
Intervention Model Description: The intervention group is compared with the control group.
Masking Description: The study is a open-label trial. The pharmacist know, whether the patient is randomized to the intervention group or the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group received the normal care following the Danish standard procedure.
- Intervention group (Active Comparator): Participants in the intervention group received the normal care following the Danish stadard procedure. Additionally the participants was also offered the possibility to contact a hospital pharmacy department by phone or mail for drug counseling.
  Interventions: Other: Drug counseling

INTERVENTIONS:
Other: Drug counseling — Participants can contact a hospital pharmacy department by phone or mail and ask questions regarding drug-related issues.
  Arms: Intervention group

SUMMARY:
Objective:

The aim of this study is to evaluate if offering drug counseling from a hospital pharmacy increases patient satisfaction and sense of security regarding drug treatment after hospital discharge.

DETAILED DESCRIPTION:
Method and design:

This study was estimated to include 250 participants in a clinical randomized controlled trial. The participants were included from the Acute Medical Ward and the Department of Respiratory Medicine at Bispebjerg Hospital when discharged. The participants were randomized to one of two groups with unequal sizes: the control (50 participants) or intervention group (200 participants). This study used blocked randomization with block sizes of 5/10/15/20/25. The control group received the normal care following the Danish standard procedure. Participants in the intervention group also received the normal care but was also offered the possibility to contact a hospital pharmacy department by phone or mail and ask questions regarding drug-related issues.

Data for the primary outcome measures was collected 14 days after discharge through structured phone interviews. An interview guide with a semi-structured questionnaire and already validated questions were developed, pre-tested and optimized. The participants were asked to answer open-ended questions, closed-ended question and rate statements or questions on a five-point scale.

The participants in the control group were asked to answer 13 items (seven questions or statements on a five-point scale, four closed-ended questions and two open-ended questions).

The participants in the intervention group who did not make any queries were asked the same questions as the participants in the control group and additionally three closed-ended questions. A total of 16 items.

The participants in the intervention group who made queries were asked the same questions as the participants in the intervention group who did not make any queries and additionally five questions on a five-point scale, four closed-ended and one open-ended question. A total of 27 items.

The effect of the drug counseling regarding patient safety was evaluated by a pharmaceutical assessment in which it was assessed whether the drug counseling had potentially prevented a drug-related problem.

Quantitative data from the phone interviews will be analyzed in Microsoft excel with descriptive statistics and simple parametric statistics. An analysis will determine whether there is a difference in the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from the acute medical ward and department of respiratory medicine at Bispebjerg Hospital.
* Patients discharged to own home.
* Can speak the danish language.
* ≥18 years old.
* Can be contacted by phone.

Exclusion Criteria:

* Cognitive and communicative problems (e.g. dementia, aphasia, suicidal) or other barriers that unable the participant to use the intervention service.
* Patient does not answer phone within five attempts on five different days, when trying to conduct patient interview.
* Cognitive and communicative problems that unable the participant to answer questions in the patient interview.
* Deceased or readmitted before patient interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Sense of security regarding drug treatment and satisfaction with drug counseling. | 2-4 weeks after discharge.
  The questionnaire comprised closed-ended questions, open-ended questions and questions or statements where the respondents were asked to rate the questions or statements on a five-point scale. The scale used is a attitude measurement scale that assess attitudes by presenting respondents with sentences that state beliefs about the particular attitude being measured. The respondents then decide to what extent he or she agrees with the statement. The responses are divided numerically into a series of ordered responses. Ratings: 1 = not at all, 2 = to a small extent, 3 = to some extent, 4 = to a great extent, 5 = to a very great extent.

SECONDARY OUTCOMES:
Number of medications by admission. | Within one week after discharge.
  Number of medications will be read in admission report.
Number of medications by discharge. | Within one week after discharge.
  Number of medications will be read in discharge report..
Number of patients that received medication review by pharmacist during admission. | Within one week after discharge.
  The patient's journal will be searched for a medication review.
Number of patients that received help with medication at home after discharge. | Within one week after discharge.
  The patient's journal will be searched for information regarding help with medication at home.
Number of enquiries. | Directly after the patient received drug counseling.
  Patient enquiries will be classified to one of the predefined categories: adverse effects, choice of therapy, dosage and administration, interactions, product information, storage and handling, indication or other.
Number of potentially prevented drug-related problems. | Directly after the patient received drug counseling.
  The pharmacist that performed the drug counseling assessed whether the drug counseling had potentially prevented a drug-related problem.
Cause of hospitalization. | Within one week after discharge.
  The patient's journal will be searched for cause of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Tim E Vejborg, M.Sc.Pharm, Principal Investigator — Region Hovedstadens Apotek
Locations (1):
- Capital Regions Hospital Pharmacy, Copenhagen, København NV, Denmark

REFERENCES:
- [Derived] Fjaere KW, Vejborg TE, Colberg L, Ulrich CS, Pedersen L, Demeny AK, Poulsen JH, Armandi HB, Clemmensen MH. Medicine information helpline after hospitalization-a randomized trial: Impact on patient satisfaction, patient concerns about medicines and clinical outcome on patient safety. PLoS One. 2023 Oct 26;18(10):e0293523. doi: 10.1371/journal.pone.0293523. eCollection 2023. PMID 37883413